CLINICAL TRIAL: NCT01839799
Title: A Randomized Phase II/Genomic Trial of Two Chemotherapy Regimens in Patients With Resected Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03213
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Patients; with; resected
MeSH Terms: interventions — Gemcitabine; Albumin-Bound Paclitaxel; Paclitaxel; folfirinox; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - FOLFIRINOX (Experimental): FOLFIRINOX:
  Irinotecan 180 mg/m2 Day 1 Oxaliplatin 85 mg/m2 Day 1 5-FU 400 mg/m2 bolus with Leucovorin 200 mg/m2 over 2h, Day 1, then 5-FU 2400 mg/m2 over 46h. Four cycles over 8 weeks
  Chemoradiation:
  Radiation to begin no sooner than 28 days from last day of chemotherapy.
  On Day 1(+ 2days to accommodate scheduling difficulties):
  Infusional 5-FU (225 mg/m2 continuous infusion during radiation) and radiation therapy as defined.
  FOLFIRINOX:
  Irinotecan 180 mg/m2 Day 1 Oxaliplatin 85 mg/m2 Day 1 5-FU 400 mg/m2 bolus with Leucovorin 200 mg/m2 over 2h, Day 1, then 5-FU 2400 mg/m2 over 46h. Four cycles, if tolerated
  Interventions: Drug: FOLFIRINOX; Radiation: Chemoradiation
- Arm 2 - Gemcitabine / Abraxane (Experimental): Gemcitabine / Abraxane Gemcitabine 1000 mg/m2 Days 1, 8, 15 Abraxane 125 mg/m2 Days 1, 8, 15 Two cycles over 8 weeks
  Chemoradiation:
  Radiation to begin no sooner than 28 days from last day of chemotherapy. On Day 1 (+ 2days to accommodate scheduling difficulties) Infusional 5-FU (225 mg/m2 continuous infusion during radiation) and radiation therapy as defined.
  Gemcitabine / Abraxane Gemcitabine 1000 mg/m2 Days 1, 8, 15 Abraxane 125 mg/m2 Days 1, 8, 15 Two cycles, if tolerated
  Interventions: Drug: Gemcitabine; Drug: Abraxane; Radiation: Chemoradiation

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 IV over 30 to 100 minutes, day 1, 8, 15
  Other Names: Gemzar
  Arms: Arm 2 - Gemcitabine / Abraxane
Drug: Abraxane — 125 mg/m2 IV over 30 minutes, day 1, 8, 15
  Other Names: Paclitaxel
  Arms: Arm 2 - Gemcitabine / Abraxane
Drug: FOLFIRINOX — Irinotecan 180 mg/m2 Day 1 Oxaliplatin 85 mg/m2 Day 1 5-FU 400 mg/m2 bolus with Leucovorin 200 mg/m2 over 2h, Day 1, then 5-FU 2400 mg/m2 over 46h. Four cycles, if tolerated
  Arms: Arm 1 - FOLFIRINOX
Radiation: Chemoradiation

SUMMARY:
Determine the relapse-free survival of resected pancreatic cancer patients following two novel regimens with activity in advanced disease.

DETAILED DESCRIPTION:
This trial is a randomized Phase II study of FOLFIRINOX versus gemcitabine/abraxane in patients with completely resected pancreatic cancer (Stages I-III). Patients will receive eight weeks of chemotherapy, then 5-FU/radiation, then another 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed evidence of pancreatic carcinoma.
* Patients must have had all gross disease resected (R0 or R1 resection, patients who underwent an R2 resection are not eligible).
* Patients must have had no prior chemotherapy or radiation therapy for pancreatic cancer.
* Age > 18 years.
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients must have normal organ and marrow function measured within 2 weeks, prior to registration as follows:

Absolute Neutrophil Count (ANC) > 1,500/µL Platelets > 100,000/µL Total bilirubin less than 2-fold upper limit of normal (ULN) Aspartate Aminotransferase (AST)/alanine aminotransferase (ALT)<2.5X institutional upper limit of normal Creatinine clearance > 60mL/min for patients with creatinine levels above institutional normal.

* Patients must be > 4 weeks and < 12 weeks post-surgery at time of study registration.
* Women of childbearing potential and sexually active males are strongly advised to use appropriate contraceptive measures.
* Women must not be pregnant or breast-feeding.

Exclusion Criteria:

* Patients receiving any other investigational agents.
* Patients with known metastases.
* Patients with wounds that have not fully healed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX: FOLFIRINOX: Irinotecan 180 mg/m2 Day 1 Oxaliplatin 85 mg/m2 Day 1 5-FU 400 mg/m2 bolus with Leucovorin 200 mg/m2 over 2h, Day 1, then 5-FU 2400 mg/m2 over 46h. Four cycles, if tolerated
  Chemoradiation
- Gemcitabine/Abraxane: Gemcitabine: 1000mg/m2 IV over 30 to 100 minutes, day 1, 8, 15
  Abraxane: 125 mg/m2 IV over 30 minutes, day 1, 8, 15
  Chemoradiation
Period: Overall Study
Arm/Group | FOLFIRINOX | Gemcitabine/Abraxane
Started | 17 | 15
Completed | 17 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine: Gemcitabine: 1000mg/m2 IV over 30 to 100 minutes, day 1, 8, 15
  Abraxane: 125 mg/m2 IV over 30 minutes, day 1, 8, 15
  Chemoradiation
- Total: Total of all reporting groups
Arm/Group | FOLFIRINOX | Gemcitabine | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 11 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse-free Survival
Description: In this small trial we will regard a median progression-free survival of 20 months as indicative of potential therapeutic benefit meriting additional study.
Time Frame: 20 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: FOLFIRINOX: Irinotecan 180 mg/m2 Day 1 Oxaliplatin 85 mg/m2 Day 1 5-FU 400 mg/m2 bolus with Leucovorin 200 mg/m2 over 2h, Day 1, then 5-FU 2400 mg/m2 over 46h. Four cycles, if tolerated
  Chemoradiation
- Arm 2: Gemcitabine: 1000mg/m2 IV over 30 to 100 minutes, day 1, 8, 15
  Abraxane: 125 mg/m2 IV over 30 minutes, day 1, 8, 15
  Chemoradiation
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 17 | 15
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 4/17 | 6/15
Other Adverse Events (participants affected / at risk) | 17/17 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=17) | Arm 2 (N=15)
Viral Syndrome (Infections and infestations) | 1 | 0
Fever (General disorders) | 4 | 1
anemia (Gastrointestinal disorders) | 1 | 0
GI Bleed (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
hepatic infection (SAE) (Infections and infestations) | 1 | 0
Non-neutropenic fever (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
increased abd distention (Metabolism and nutrition disorders) | 1 | 0
Abdominal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bacteremia-E.Coli (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Chills (General disorders) | 0 | 1
decrease wbc (Investigations) | 2 | 0
decreased neutrophils (Investigations) | 1 | 0
protein malnutrition (Metabolism and nutrition disorders) | 1 | 0
decreased appetite (Metabolism and nutrition disorders) | 1 | 0
CMV (Infections and infestations) | 1 | 0
Septic Shock (Gastrointestinal disorders) | 0 | 1
Bilatteral Hip Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fever /+ blood culture (General disorders) | 0 | 1
SmBowel Obstruction (Gastrointestinal disorders) | 0 | 1
PRESS (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=17) | Arm 2 (N=15)
nausea (Gastrointestinal disorders) | 13 | 5
fatigue (General disorders) | 14 | 13
anemia (Blood and lymphatic system disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 14 | 7
rash (Skin and subcutaneous tissue disorders) | 3 | 4
elevated ALK Phos (Investigations) | 1 | 0
anorexia (Metabolism and nutrition disorders) | 3 | 1
elevated creatinine (Investigations) | 0 | 0
elevated trigylcerides (Investigations) | 0 | 0
thrombocytopenia (Investigations) | 1 | 1
elevated ALT (Investigations) | 0 | 4
headache (Nervous system disorders) | 1 | 1
hyperkalemia (Investigations) | 0 | 0
mucositis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 10 | 3
dry mouth (Gastrointestinal disorders) | 0 | 0
dysgeusia (Nervous system disorders) | 2 | 1
edema (General disorders) | 0 | 6
elevated cholesterol (Investigations) | 0 | 0
hypoalbuminemia (Investigations) | 2 | 0
pruritis (Skin and subcutaneous tissue disorders) | 0 | 0
weight loss (Investigations) | 3 | 1
blurred vision (Eye disorders) | 0 | 0
constipation (Gastrointestinal disorders) | 4 | 3
hyperglycemia (Investigations) | 4 | 0
hypokalemia (Investigations) | 5 | 1
hyponatremia (Investigations) | 0 | 0
neutropenia (Investigations) | 10 | 10
decreased wbc (Investigations) | 5 | 4
hypomagnesium (Investigations) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 6 | 0
skin infection port (Skin and subcutaneous tissue disorders) | 1 | 0
abd/cramping/pain (Musculoskeletal and connective tissue disorders) | 1 | 1
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
peripheral neuropathy (Nervous system disorders) | 2 | 1
Dizziness (General disorders) | 2 | 0
Decreased Platlets (Investigations) | 3 | 1
Ear Bleed -L-ear (Ear and labyrinth disorders) | 1 | 0
increased Ast (Investigations) | 1 | 0
decreased plt (Investigations) | 3 | 1
hypotension (Investigations) | 2 | 2
Insomnia (Psychiatric disorders) | 3 | 1
neuropathy (Nervous system disorders) | 7 | 4
loose stools/intermittent (Gastrointestinal disorders) | 1 | 2
Runny nose (Skin and subcutaneous tissue disorders) | 1 | 0
Mouth Sores (Skin and subcutaneous tissue disorders) | 6 | 1
fever (General disorders) | 5 | 4
gout (General disorders) | 1 | 0
decreased neutrophils (Investigations) | 3 | 0
protein malnutrition (Investigations) | 1 | 0
decrease wbc (Investigations) | 1 | 4
Lightheadeness (General disorders) | 1 | 0
UTI (Renal and urinary disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 6
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Myalgia (Eye disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Decreased Appetite (Investigations) | 2 | 1
Loose bowel movement (Gastrointestinal disorders) | 1 | 0
gas (Gastrointestinal disorders) | 5 | 6
abdominal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
night sweats (General disorders) | 1 | 0
flatulance (Gastrointestinal disorders) | 1 | 4
ratiation dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
hypersensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
abdominal cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Thick feeling tongue (Musculoskeletal and connective tissue disorders) | 1 | 0
paronychia (Infections and infestations) | 1 | 0
Cold Sensitivity (General disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tunnel Vision (Eye disorders) | 1 | 0
Chest Pressure/Spasm (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft nails (Skin and subcutaneous tissue disorders) | 0 | 1
folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
siatica (Nervous system disorders) | 0 | 1
stomach virus (Gastrointestinal disorders) | 0 | 2
elevated AST (Investigations) | 0 | 6
malabsorption (Metabolism and nutrition disorders) | 0 | 1
orthostatic (General disorders) | 0 | 1
Flu like symptoms (General disorders) | 0 | 3
Horseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fever Other (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT01839799/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT01839799/Prot_SAP_001.pdf